CLINICAL TRIAL: NCT05622526
Title: Randomized, Double-blind, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of Fecal Microbiota Transfer by Capsules vs. Placebo for the Treatment of Patients With Nonalcoholic Steatohepatitis
Brief Title: Evaluate the Efficacy, Safety and Tolerability of Fecal Microbiota Transfer for the Treatment of Patients With Nonalcoholic Steatohepatitis
Acronym: EMOTION
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMOTION
Record Dates: First submitted 2022-09-21; First posted 2022-11-18 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Patients With Nonalcoholic Steatohepatitis
Keywords: MetEH: metabolic hepatic steatosis; NASH nonalcoholic steatohepatitis; TMF: fecal microbiota transplantation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 or Experimental group (Experimental): treatment with an initial dose of 24 oral capsules of MBK-01 and a maintenance dose of 12 oral capsules of MBK-01 every 3 months (4 maintenance doses).
  Interventions: Drug: Group 1 or Experimental group
- Group 2 or Control group (Placebo Comparator): treatment with an initial dose of 24 oral capsules of MBK-01 and a maintenance dose of 12 oral capsules of MBK-01 every 3 months for 12 months (4 maintenance doses)
  Interventions: Other: Group 2 or Control group

INTERVENTIONS:
Drug: Group 1 or Experimental group — Capsules of fecal microbiota transplantation
  Arms: Group 1 or Experimental group
Other: Group 2 or Control group — capsules of placebo
  Arms: Group 2 or Control group

SUMMARY:
The EMOTION study is a multicentric, double-blind, controlled, parallel-group, phase IIa randomized Clinical trial to evaluate the efficacy, safety and tolerability of TMF capsules for the treatment of patients with NASH.

The clinical trial has two stages:

* Screening phase with a duration of 12 weeks to classify patients based on lifestyle modifications.
* Treatment phase where patients will be randomized and stratified 2:1 to treatment:
* Experimental for n=64 patients.
* Placebo control for n=32 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders aged between 18 and75 years old (both included).
2. Body mass index (BMI) <40 kg/m2.
3. Histological diagnosis of NASH, accepted by EASL and AASLD , from a liver biopsy obtained up to 24 weeks prior to the signing of the informed consent.
4. NASH histologic activity score (NAS) ≥ 4, with a score of 1 or more in each subcomponent (steatosis, lobular inflammation, and liver cell ballooning).
5. Histologic evidence of stage 1 fibrosis (with perisinusoidal or portal fibrosis), stage 2 (perisinusoidal and portal/periportal fibrosis), or stage 3 (bridging fibrosis) as defined by the NASH CRN fibrosis score.

Exclusion Criteria:

1. Evidence of other type of liver disease.
2. History of high alcohol intake (daily consumption > 30 g/day for men and > 20 g/day for women).
3. Weight change of more than 5% in the 3 months prior to screening.
4. Subjects with HbA1c> 9.5%. For subjects with an HbA1c> 9.5% at the screening visit, a repeat test may be performed within the screening window.

   A repeated result of HbA1c> 9.5% will result in exclusion.
5. Diabetic patients with:

   * Insulin treatment.
   * Changes in antidiabetic medication in the 4 months prior to liver biopsy according to the following conditions:
   * Modification of the dose of treatment with glucagon agonists type 1 (GLP-1).
   * Implementation of treatment with a new antidiabetic.
6. History of bariatric surgery.
7. Cirrhosis.
8. Portal thrombosis.
9. Known or suspected hepatocellular carcinoma.
10. Clinically significant gastrointestinal, cardiovascular, neurological, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory or infectious disease, as determined by the investigator.
11. An estimated glomerular filtration rate (eGFR) <45 ml / min / 1.73 m2 (calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] method).
12. Medical conditions that decrease life expectancy to less than 2 years, including cancer.
13. Presence of an inherited or acquired immunodeficiency.
14. Diagnosis of inflammatory bowel disease (Crohn's disease, ulcerative colitis, microscopic colitis), active irritable bowel syndrome (within the last 2 years according to Rome IV criteria), celiac disease not well controlled with a gluten-free diet, active gastroparesis, toxic megacolon.
15. Major intra-abdominal surgery in the 2 months prior to randomization of the patient in the study.
16. Antibiotic intake in the 8 weeks prior to the screening date.
17. Probiotic/prebiotic/marketed synbiotic intake in the 4 weeks prior to the screening date.
18. Pregnancy or lactation.
19. Any other condition that, in the opinion of the investigator, could prevent or hinder compliance.
20. Use of medication with potential steatogenic effect (corticosteroids, valproic acid, amiodarone and/or tamoxifen) within the 6 months prior to the first dose of study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with improvement of fat fraction by proton density by MRI and no worsening of activity or fibrosis. | 72 weeks
number of adverse events (AEs), serious AEs, AEs resulting in discontinuation of study treatment, AEs of special interest, and changes in vital signs and laboratory values | 72 weeks

SECONDARY OUTCOMES:
Proportion of patients with improvement (at least one point) in lobular swelling and/or ballooning without worsening of fibrosis. | 72 weeks
NAFLD Fibrosis score | 72 weeks
Changes in weight, BMI. | 72 weeks
Changes in systolic and diastolic blood pressure, lipid profile, carotid ultrasound. | 72 weeks
Changes in the quality of life questionnaire specific to chronic liver disease due to NAFLD. | 72 weeks
patient-reported outcomes | 72 weeks